CLINICAL TRIAL: NCT05001711
Title: Acute Feasibility Study Assessing Safety and Performance of Aria CV Acute PH System in Patients With WHO Group 2 and 3 Pulmonary Hypertension
Brief Title: Acute Assessment of the Aria CV System in Patients With WHO Groups 2 and 3 Pulmonary Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aria CV, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARIACV202101
Record Dates: First submitted 2021-07-26; First posted 2021-08-12 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WHO Group 2 (Experimental)
  Interventions: Device: Aria CV Acute PH System
- WHO Group 3 (Experimental)
  Interventions: Device: Aria CV Acute PH System

INTERVENTIONS:
Device: Aria CV Acute PH System — The Aria CV Acute PH System is indicated for evaluation of hemodynamic responses (e.g. pulmonary arterial compliance, cardiac output, and effective arterial elastance) to an intravascular Balloon catheter temporarily placed in the pulmonary artery in symptomatic adult patients with WHO Group 2 or WHO Group 3 pulmonary hypertension and right ventricular dysfunction.

SUMMARY:
This study is a prospective, non-randomized, two arm, single-center acute feasibility study assessing safety and performance of the Aria CV Acute PH System in WHO Group 2 and 3 PH patients.

DETAILED DESCRIPTION:
This study is a prospective, non-randomized, two arm, single-center acute feasibility study assessing safety and performance of the Aria CV Acute PH System in WHO Group 2 and 3 PH patients.

The planned enrollment is a maximum enrollment of 40 patients to ensure up to 10 "Device Deployed" subjects in each arm at one site.

The duration of study participation for each subject is expected to be approximately 60 days.

ELIGIBILITY:
Inclusion Criteria for WHO Group 2

1. 18 years or older
2. Symptomatic WHO Functional Class (FC) III
3. Based on preexisting echocardiography within the past 6 months, evidence of right heart dysfunction: RV ejection fraction (RVEF) < 45% by visual estimate, and at least one of the following:

   1. Tricuspid Annulus Plane Systolic Excursion (TAPSE) ≤16 mm
   2. RV Fractional area change <35%
   3. RVs' velocity < 10 cm/s
   4. RV free wall strain <18%
   5. RVEF < 35% by visual estimate
4. MPA diameter > 32mm and length >70 mm as determined by preexisting fluoroscopy, echocardiography, computerized tomography, or magnetic resonance imaging within the past 6 months.
5. Elevated pulmonary arterial pressure based on preexisting resting RHC within the past 6 months: Mean PAP (mPAP) > 30 mmHg
6. Intra-procedural confirmation of elevated pulmonary arterial pressure based on resting RHC: mPAP > 30 mmHg
7. Patient is willing and able to provide informed consent.
8. Previous diagnosis of left heart dysfunction.
9. Intra-procedural confirmation of WHO Group 2 diagnosis based on resting RHC:

   1. PAWP: >15 and ≤30 mmHg, and
   2. Combined post- and pre-capillary pulmonary hypertension (CpcPH), defined as PVR > 3 WU

Exclusion Criteria for WHO Group 2

1. Anatomy not suitable for RHC
2. Anatomy not suitable for placement of Aria CV Acute Device:

   1. Contraindication to 16 Fr femoral vein access
   2. Body habitus that would preclude safe placement of any components of Aria CV Acute Device
3. Any previous tricuspid valvular surgery, percutaneous valve repair, or presence of prosthetic cardiac device such as pacemaker or defibrillator leads, or vena cava filter that in the opinion of the investigator may interfere with investigational device placement or performance
4. Uncontrolled atrial fibrillation
5. Sustained tachyarrhythmia (heart rate >110/min) at time of index procedure
6. Right heart valve regurgitation:

   1. Moderate to severe (Grade 3 or 4) pulmonary valve regurgitation
   2. Severe (Grade 4) tricuspid valve regurgitation
7. Patient with any of the following medical history or comorbidities:

   1. History of unprovoked Pulmonary Embolism or CTEPH
   2. Currently on dialysis
   3. Current or recent (<6 months prior to planned index procedure) endocarditis
   4. Clinically significant patent foramen ovale or other inter-atrial or inter-ventricular shunt
   5. Current active systemic infection requiring antibiotic therapy
8. As determined by the physician the subject is medically unstable and/or represents an unreasonable procedural risk.
9. Hypersensitivity or contraindication to

   1. Required medications (e.g. contrast agents, heparin) which cannot be adequately managed, or
   2. Materials in investigational device including polyurethane, silicone, nickel, and titanium
10. Pregnant or lactating woman
11. Currently participating in other investigational drug or device trials that may interfere with the outcome of this study
12. Diagnosis of WHO Groups 1, 3, 4 or 5 PH
13. Previous diagnosis of idiopathic hypertrophic subaortic stenosis (IHSS, also known as hypertrophic obstructive cardiomyopathy-HOCM)
14. Untreated aortic or mitral stenosis

Inclusion Criteria for WHO Group 3

1. 18 years or older
2. Symptomatic WHO Functional Class (FC) III
3. Based on preexisting echocardiography within the past 6 months, evidence of right heart dysfunction: RV ejection fraction (RVEF) < 45% by visual estimate, and at least one of the following:

   1. Tricuspid Annulus Plane Systolic Excursion (TAPSE) ≤16 mm
   2. RV Fractional area change <35%
   3. RVs' velocity < 10 cm/s
   4. RV free wall strain <18%
   5. RVEF < 35% by visual estimate
4. MPA diameter > 32mm and length >70 mm as determined by preexisting fluoroscopy, echocardiography, computerized tomography, or magnetic resonance imaging within the past 6 months
5. Elevated pulmonary arterial pressure based on preexisting resting RHC within the past 6 months: Mean PAP (mPAP) > 30 mmHg
6. Intra-procedural confirmation of elevated pulmonary arterial pressure based on resting RHC: mPAP > 30 mmHg
7. Patient is willing and able to provide informed consent
8. Previous diagnosis of chronic obstructive pulmonary disease (COPD) or interstitial lung disease (ILD) including idiopathic pulmonary fibrosis (IPF) or combined emphysema with fibrosis
9. Intra-procedural confirmation of WHO Group 3 diagnosis based on resting RHC:

   1. PAWP≤ 15 mmHg, and
   2. PVR > 4 WU

Exclusion Criteria for WHO Group 3

1. Anatomy not suitable for RHC
2. Anatomy not suitable for placement of Aria CV Acute Device:

   1. Contraindication to 16 Fr femoral vein access
   2. Body habitus that would preclude safe placement of any components of Aria CV Acute device
3. Any previous tricuspid valvular surgery, percutaneous valve repair, or presence of prosthetic cardiac device such as pacemaker or defibrillator leads, or vena cava filter that in the opinion of the investigator may interfere with investigational device placement or performance
4. Uncontrolled atrial fibrillation
5. Sustained tachyarrhythmia (heart rate >110/min) at time of index procedure
6. Right heart valve regurgitation:

   1. Moderate to severe (Grade 3 or 4) pulmonary valve regurgitation
   2. Severe (Grade 4) tricuspid valve regurgitation
7. Patient with any of the following medical history or comorbidities:

   1. History of unprovoked Pulmonary Embolism or CTEPH
   2. Currently on dialysis
   3. Current or recent (<6 months prior to planned index procedure) endocarditis
   4. Clinically significant shunt such as patent foramen ovale, inter-atrial or inter-ventricular shunt, or other.
   5. Current active systemic infection requiring antibiotic therapy
8. As determined by the physician the subject is medically unstable and/or represents an unreasonable procedural risk.
9. Hypersensitivity or contraindication to

   1. Required medications (e.g. contrast agents, warfarin, heparin) which cannot be adequately managed, or
   2. Materials in investigational device including polyurethane, silicone, nickel, and titanium.
10. Pregnant or lactating woman
11. Currently participating in other investigational drug or device trials that may interfere with the outcome of this study
12. Diagnosis of WHO Groups 1, 2, 4 or 5 PH

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-01-06 (Actual)

PRIMARY OUTCOMES:
Primary Safety Endpoint | 30 Days
  Incidence of investigational device-related serious adverse events (SAEs) through 30 days post-index procedure, based on Clinical Events Committee assessment.

SECONDARY OUTCOMES:
Secondary Safety Endpoint | 30 Days
  All reported adverse events occurring during the study will be summarized by the CEC for seriousness and relatedness based on site-reported data.

CONTACTS AND LOCATIONS:
Overall Officials: Irene M Lang, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria